CLINICAL TRIAL: NCT03641807
Title: The Comparison of Three Different Modes of Assessment on Acupuncture Effect on Patients With Chronic Prostatitis/Chronic Pelvic Pain Syndrome: a Study Protocol for a Randomized Controlled Trial
Brief Title: Different Modes of Assessment on Acupuncture Effect on Patients With Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhou Jing, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-098-KY
Record Dates: First submitted 2018-08-14; First posted 2018-08-22 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Chronic Prostatitis; Chronic Pelvic Pain Syndrome
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental)
  Interventions: Other: Acupuncture
- Sham acupuncture (Sham Comparator)
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Acupuncture — Bilateral BL23, BL33, BL35 and SP6 will be inserted using Hwato-brand disposable acupuncture needles. With patients prone, after routine sterilization, bilateralBL33 will be inserted to a depth of 50 to 60mm with a 30° to 45° angle in an inferomedial direction using needles (0.30mm in diameter, 75mm in length). Bilateral BL35 will be inserted to a depth of 50 to 60mm with a slightly superolateral direction using needles (0.30mm in diameter, 75mm in length). BL23 and SP6 will be inserted vertically to a depth of 25 to 30mm using needles (0.30mm in diameter, 40mm in length). Manipulation of the needles by lifting and thrusting combined with twirling and rotating evenly will be performed until deqi occurs, defined as a sensation of soreness, numbness, heaviness, and ache. Manipulations will be applied every 10minutes and each session will last for 30minutes.
  Arms: Acupuncture
Other: Sham acupuncture — Bilateral sham BL 23, BL 33, BL 35 (15mmto BL23, BL33, and BL35) and SP6 (10mmto SP6) will be inserted by needles (0.20mm in diameter, 25mm in length) to a depth of 2 to 3mm without manipulation.
  Arms: Sham acupuncture

SUMMARY:
Background: Chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) is a common disorder. Some studies have indicated that acupuncture may ameliorate the symptoms of CP/CPPS. However, results are varied and range widely, perhaps due to different modes of assessment including timepoints, places of assessment, and especially subjective scales. We propose to determine the efficacy of acupuncture relative to sham acupuncture for patients with CP/CPPS, and compare different modes of assessment regarding the therapeutic effects of acupuncture.

Methods: Sixty patients with CP/CPPS will be randomly assigned to receive either acupuncture or sham-acupuncture (30 patients, each). Treatment will be conducted 3 times/week, for 4 weeks. The primary outcomes will each be the change from baseline of the total NIH (National Institutes of Health) CPSI (Chronic Prostatitis Symptom Index) score associated with 3 modes of assessment: Mode 1, the scale recorded at the hospital within 10minutes after the last session of 4 weeks of acupuncture treatment, in the company of the outcome assessors; Mode 2, the scale recorded the same day, but not at the hospital; and Mode 3, the scale recorded at the hospital 1 to 3 days after the last acupuncture session. The 3 key secondary outcomes include will be the 3 modes assessment of the changes from baseline of the NIH-CPSI total scores in the acupuncture group at week 4 after treatment. Analysis was by intention-to-treat, and multiplicity was controlled for with a step-down closed-testing procedure.

ELIGIBILITY:
Inclusion Criteria:

* meet the diagnostic criteria according to the NIH CP/CPPS consensus: discomfort or pain in the pelvic region for at least 3 months in the previous 6 months
* 18-50 years
* NIH-CPSI total score ≥15

Exclusion Criteria:

* Urologic disease
* Residual urine volume ≥100 milliliter (mL)
* Qmax ≤15mL/s
* Use 5-alpha reductase inhibitor, alpha-blockers, antibiotics or any other prostatitis-specific medication during previous 1 month
* Diseases that influence urologic symptoms are multiple sclerosis, multiple system atrophy, stroke, Alzheimer disease, Parkinson's disease, spinal cord injury, cauda equina injury, and sexually transmitted disease
* Any acute disease or severe disease requiring treatment

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in total score of National Institutes of Health-chronic prostatitis symptom index (NIH-CPSI) measured by the assessment of mode 1 | week 4
  The National Institutes of Health-chronic prostatitis symptom index (NIH-CPSI) has a total score range from 0 to 43 and higher scores indicate more severe symptoms. The 9 items of this scale are stratified into 3 domains which are pain/discomfort (location/type, frequency and severity, 0-21 points), urinary symptoms (10 points) and quality of life (0-12 points). Mode 1, the scale is recorded at the hospital within 10minutes after the twelfth (last) treatment of the 4-week treatment period, in the company of the outcome assessors.
The change from baseline in total score of National Institutes of Health-chronic prostatitis symptom index (NIH-CPSI) measured by the assessment of mode 2 | week 4
  The National Institutes of Health-chronic prostatitis symptom index (NIH-CPSI) has a total score range from 0 to 43 and higher scores indicate more severe symptoms. The 9 items of this scale are stratified into 3 domains which are pain/discomfort (location/type, frequency and severity, 0-21 points), urinary symptoms (10 points) and quality of life (0-12 points). Mode 2, the scale is recorded the same day, but not at the hospital.
The change from baseline in total score of National Institutes of Health-chronic prostatitis symptom index (NIH-CPSI) measured by the assessment of mode 3 | 1 to 3 days after the last acupuncture session
  The National Institutes of Health-chronic prostatitis symptom index (NIH-CPSI) has a total score range from 0 to 43 and higher scores indicate more severe symptoms. The 9 items of this scale are stratified into 3 domains which are pain/discomfort (location/type, frequency and severity, 0-21 points), urinary symptoms (10 points) and quality of life (0-12 points). Mode 3, the scale is recorded at the hospital 1 to 3 days after the last acupuncture session.

SECONDARY OUTCOMES:
Mode 1 of assessment of the changes from baseline of NIH-CPSI total score in the acupuncture group | week 4
  The National Institutes of Health-chronic prostatitis symptom index (NIH-CPSI) has a total score range from 0 to 43 and higher scores indicate more severe symptoms. The 9 items of this scale are stratified into 3 domains which are pain/discomfort (location/type, frequency and severity, 0-21 points), urinary symptoms (10 points) and quality of life (0-12 points). Mode 1, the scale is recorded at the hospital within 10minutes after the twelfth (last) treatment of the 4-week treatment period, in the company of the outcome assessors.
Mode 2 of assessment of the changes from baseline of NIH-CPSI total score in the acupuncture group | week 4
  The National Institutes of Health-chronic prostatitis symptom index (NIH-CPSI) has a total score range from 0 to 43 and higher scores indicate more severe symptoms. The 9 items of this scale are stratified into 3 domains which are pain/discomfort (location/type, frequency and severity, 0-21 points), urinary symptoms (10 points) and quality of life (0-12 points). Mode 2, the scale is recorded the same day, but not at the hospital.
Mode 3 of assessment of the changes from baseline of NIH-CPSI total score in the acupuncture group | 1 to 3 days after the last acupuncture session
  The National Institutes of Health-chronic prostatitis symptom index (NIH-CPSI) has a total score range from 0 to 43 and higher scores indicate more severe symptoms. The 9 items of this scale are stratified into 3 domains which are pain/discomfort (location/type, frequency and severity, 0-21 points), urinary symptoms (10 points) and quality of life (0-12 points). Mode 3, the scale is recorded at the hospital 1 to 3 days after the last acupuncture session.
The change from baseline of subscales scores of NIH-CPSI | week 4
  The National Institutes of Health-chronic prostatitis symptom index (NIH-CPSI) has a total score range from 0 to 43 and higher scores indicate more severe symptoms. The 9 items of this scale are stratified into 3 domains which are pain/discomfort (location/type, frequency and severity, 0-21 points), urinary symptoms (10 points) and quality of life (0-12 points).
The change from baseline of International Prostate Symptom Score (IPSS) | week 4
  International Prostate Symptom Score (IPSS) (Hong Kong Chinese version 2) is a valid, reliable and sensitive measure to assess Chinese males with 7 questions concerning urinary symptoms and 1 question concerning quality of life [34]. Total score of IPSS ranges from 0-35 (asymptomatic to very symptomatic). Symptoms evaluated by IPSS are categorized as mild (0-7), moderate (8-19) and severe (20-35).
The proportions of participants in each response category of the Global Response Assessment (GRA) | week 4
  Global Response Assessment (GRA) which is composed of 7 response categories: markedly worsened, moderately worsened, slightly worsened, no change, slightly improved, moderately improved, and markedly improved.

OTHER OUTCOMES:
Expectancy of acupuncture | Baseline
  Participants need to answer two questions: "In general, do you believe acupuncture is effective for treating the illness?" and "Do you think acupuncture will be helpful to improve your CP/CPPS symptoms?" Participants will choose "Unclear", "Yes" or "No" as the answer.
Blinding assessment | week 4
  Participants will be asked to reply to the question ("Do you think you have received traditional acupuncture in the past weeks?") after treatment (sessions 11 or 12) within 5 minutes. The participants will be able to choose one of the following options as the answer: "Unclear", "Yes" or "No".
Incidence of adverse events (AEs) related with acupuncture | week 1 to week 4
  AEs related to acupuncture include severe pain (assessed by VAS, 7 points at least), broken needle, fainting, local hematoma, localized infection and post-acupuncture discomfortable symptoms such as nausea, vomiting, palpitation, dizziness, headache, anorexia and insomnia, etc. during treatment period.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The First Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - Hengyang Hospital Affiliated to Hunan University of Chinese Medicine, Hengyang, Hunan
  - Yantai Hospital of Traditional Chinese Medicine, Yantai, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan